CLINICAL TRIAL: NCT04505982
Title: Anti IL6R Reduce Complement Serum Level in Rheumatoid Arthritis Patients: Facts and Implications: Monocentric Study in Belgian Center
Brief Title: Anti IL6R Reduce Complement Serum Level in Rheumatoid Arthritis Patients: Facts and Implications
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BADOT, Valerie (Other)
Responsible Party: Sponsor-Investigator, BADOT, Valerie, Head of rhumatology department, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-IL6
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Rheumatoid Polyarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Tocilizumab intravenous: Patients followed in the CHU Brugmann Hospital for a rheumatoid polyarthritis and treated according to standard of care with tocilizumab, intravenous
  Interventions: Other: Data extraction from medical files
- Tocilizumab subcutaneous: Patients followed in the CHU Brugmann Hospital for a rheumatoid polyarthritis and treated according to standard of care with tocilizumab, subcutaneous
  Interventions: Other: Data extraction from medical files
- Sarilumab subcutaneous: Patients followed in the CHU Brugmann Hospital for a rheumatoid polyarthritis and treated according to standard of care with sarilumab, subcutaneous
  Interventions: Other: Data extraction from medical files

INTERVENTIONS:
Other: Data extraction from medical files — Data extraction from medical files

SUMMARY:
Interleukin 6 is identified as a cytokine with pro and anti-inflammatory effects, depending on the context to which it is exposed, exerting a role in the expansion and activation of T lymphocytes, in the survival, expansion and the maturation of B lymphocytes and plasmablasts as well as in the regulation of the acute phase response. The IL-6 receptor complex is a dimer in which each monomer is composed of an 80 kD subunit, IL-6R or CD126, expressed in hepatocytes, leukocytes and in megakaryocytes, which binds IL- 6 and a 130 kD subunit, gp130 or CD130, which is expressed ubiquitously. Its effects are mediated mainly by the way of tyrosine kinases of the Jaks family, and transcription factors of the STATs family.

The complement system is made up of a set of plasma proteins, cascading through three activation pathways (classical, alternate and lectin pathway). This system is considered part of innate immunity. It is also part of the acute phase response.The complement has several functions: cell lysis by formation of the membrane attack complex; opsonization and activation of phagocytosis of foreign particles, elimination of circulating immune complexes, and regulation of the adaptive immunity response and inflammation via anaphylatoxins.

After reviewing the literature, the link between IL6 and the complement system can be summarized as an induction of factor C3 and factor B, but also probably CD55 (DAF or Decay acceleration factor) and CD59 (MAC-IP or MAC-Inhibitory Protein) by interleukin-6. The effects of IL-6 on the lectin pathway, on the other hand, seem contradictory: inhibition or induction of the synthesis of MASP1 / 3 and 2 depending on the experimental model.

It has become common knowledge that anti-IL6 receptor monoclonal antibodies, used in the treatment of patients with rheumatoid arthritis and other inflammatory conditions, reduce the serum levels of acute phase proteins and in particular the levels of CRP. But what about other acute phase proteins and in particular the complement ?

A recent study showed that the serum levels of the complement components C3 and C4 were also reduced after the use of tocilizumab and this as early as 4 weeks after the first administration. To the investigator's knowledge, this is the only study reporting a decrease in complement during treatment with anti-IL6R.

This study would allow the evaluation of complement parameters in the population of patients under treatment with antiIL6R (tocilizumab or sarilumab) within the CHU Brugmann Hospital in order to

* confirm or not this observation
* look for a possible secondary clinical consequence
* compare this decrease with the activity of the disease in order to see if it could be a marker of effectiveness
* put this decrease in parallel with the side effects / tolerance of the treatment in order to see if it could be a marker of toxicity / safety

This study will also investigate the subpopulations of B lymphocytes (memory B, transitional B, and plasmablasts) in order to assess whether the evolution of one of these lines would be predictive of a therapeutic response.

Secondly, this study would eventually allow

* to improve the understanding of the mechanisms of action of the treatment on inflammatory markers by evaluating the activity of the residual complement
* to raise the need to find new parameters for monitoring inflammatory activity in these patients, since CRP assays are not very helpful.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Regular follow-up at CHU Brugmann Hospital for confirmed rheumatoid arthritis and meeting the ACR 2010 criteria
* On tocilizumab / sarilumab or for which this treatment is about to be initiated, in intravenous or subcutaneous form

Exclusion Criteria:

* Patients with a known complement deficiency before their rheumatic pathology
* Patient with hepatic impairment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients followed in the CHU Brugmann Hospital for a rhumatoid polyarthiritis and treated according to standard of care with tocilizumab / sarilumab or for which this treatment is about to be initiated, in intravenous or subcutaneous form
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Demographic data | 5 minutes
  Age, sex
Body Mass Index | 5 minutes
  Body Mass Index
Medical History (descriptive listing) | 5 minutes
  Medical History (descriptive listing)
Neoplasia | 5 minutes
  Active neoplasia, or neoplasia dated less than 5 years
Disease Activity Score Calculator for Rheumatoid Arthritis- DAS28VS | 5 minutes
  The DAS28 is a measure of disease activity in rheumatoid arthritis . DAS stands for 'disease activity score' and the number 28 refers to the 28 joints that are examined in this assessment. A DAS28 of greater than 5.1 implies active disease, less than 3.2 low disease activity, and less than 2.6 remission.
Disease Activity Score Calculator for Rheumatoid Arthritis- DAS28CRP | 5 minutes
  The DAS28 is a measure of disease activity in rheumatoid arthritis . DAS stands for 'disease activity score' and the number 28 refers to the 28 joints that are examined in this assessment. A DAS28 of greater than 5.1 implies active disease, less than 3.2 low disease activity, and less than 2.6 remission.
Health Assessment Questionnaire (HAQ) | 5 minutes
  The Health Assessment Questionnaire Disability Index (HAQ) is developed for the assessment of disability in patients with Rheumatoid Arthritis. It focuses on two dimensions of health status, physical disability (eight categories), and pain. The eight categories review a total of 20 specific functions and evaluate patient's difficulty with activities of daily living over the past week.
Concomitant medication (descriptive listing) | 5 minutes
  Concomitant medication (descriptive listing)
Adverse events linked to the medication (descriptive listing) | 5 minutes
  Adverse events linked to the medication (descriptive listing)
Hemogram: normal (yes/no) | 5 minutes
  A hemogram contains all of the pertinent information required for assessment of hematopoiesis as well as a visual assessment of plasma appearance and measurement of total solids (an estimate of total protein) in plasma.
Leukocyte count | 5 minutes
  Leukocyte count
Blood Ionogram: normal (yes/no) | 5 minutes
  The blood ionogram analyses the ionic composition of the blood
Renal function: normal (yes/no) | 5 minutes
  Renal function
Hepatic function: normal (yes/no) | 5 minutes
  Hepatic function
Parathyroid hormone count | 5 minutes
  Parathyroid hormone count
Vitamin D count | 5 minutes
  Vitamin D count
Lipid balance: normal (yes/no) | 5 minutes
  Lipid balance allows monitoring of cholesterol (LDL-cholesterol and HDL-cholesterol) and triglycerides
Glucose concentration in the blood | 5 minutes
  Glucose concentration in the blood
Rheumatoid factor concentration | 5 minutes
  Rheumatoid factor is an autoantibody that induces inflammation and damage to the joints.
AntiCCP antibodies count | 5 minutes
  The detection of anti-CCP antibodies is used to help diagnose and prognosticate rheumatoid arthritis and differentiate it from other types of arthritis
FAN count | 5 minutes
  FAN are autoantibodies against elements of the nucleus
Sedimentation rate | 5 minutes
  Sedimentation rate
CRP count | 5 minutes
  CRP count
Complement fraction C1q count | 5 minutes
  Complement fraction C1q count
Complement fraction C3 count | 5 minutes
  Complement fraction C3 count
Complement fraction C3d count | 5 minutes
  Complement fraction C3d count
Complement fraction C3a count | 5 minutes
  Complement fraction C3a count
Complement fraction C4 count | 5 minutes
  Complement fraction C4 count
Complement fraction C4a count | 5 minutes
  Complement fraction C4a count
Complement fraction CH50 count | 5 minutes
  Complement fraction CH50 count
Complement fraction FB count | 5 minutes
  Complement fraction FB count
Lectin count | 5 minutes
  Lectin count
Lectin complement pathway serine protease 2 (MASP-2) count | 5 minutes
  Lectin complement pathway serine protease 2 (MASP-2) count
Mannose Binding lectin (MBL) count | 5 minutes
  Mannose Binding lectin (MBL) count
Complement SC5b9 count | 5 minutes
  Complement SC5b9 count
Fibrinogen count | 5 minutes
  Fibrinogen count
Lymphocyte B count: memory cells | 5 minutes
  Lymphocyte B count: memory cells
Lymphocyte B count: transitional cells | 5 minutes
  Lymphocyte B count: transitional cells
Lymphocyte B count: plasmablast cells | 5 minutes
  Lymphocyte B count: plasmablast cells

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Vandergraesen, MD, Principal Investigator — CHU Brugmann
Locations (1):
- Brugmann University Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No